CLINICAL TRIAL: NCT06281782
Title: Platelet-rich Plasma With Topical Retinoids Versus Topical Retinoids Alone in Acne Vulgaris: Randomized Clinical Trial
Brief Title: Platelet-rich Plasma With Topical Retinoids Versus Topical Retinoids Alone in Acne Vulgaris
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Howida Omar Twisy, principal investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PRP with topical retinoids
Record Dates: First submitted 2024-01-29; First posted 2024-02-28 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris | interventions — Retinoids

STUDY DESIGN:
Intervention Model Description: Topical retinoids versus topical retinoids wit PRP in acne vulgaris treatment
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topical retinoid and platelet-rich plasma (PRP) group (Active Comparator)
  Interventions: Other: topical retinoids and platalet rich plasma
- topical retinoid group (Active Comparator)
  Interventions: Other: topical retinoids and platalet rich plasma

INTERVENTIONS:
Other: topical retinoids and platalet rich plasma — We will analyse both monotherapy with a topical retinoid alone and combination therapy with a topical retinoid and platelet-rich plasma (PRP) to elucidate their role in acne treatment and provide possible recommendations for their use.

SUMMARY:
Acne vulgaris is the most common skin disease in adolescents and young adults. Adult or post-adolescent acne occurs in 12-14% of this population.It is a chronic, inflammatory disease of the pilosebaceous unit .The clinical features of acne include seborrhoea, non-inflammatory lesions (open and closed comedones), inflammatory lesions (papules and pustules), and various degrees of scarring.

Platelet-rich plasma (PRP) is prepared by simple centrifugation of whole blood to concentrate platelets and simultaneously remove red blood cells. The resultant supernatant is the PRP that contains various growth factors, including platelet-derived growth factor (PDGF), transforming growth factor (TGF), fibroblast growth factor (FGF), vascular endothelial growth factor (VEGF), and hepatocyte growth factor (HGF).These growth factors are involved in the healing of soft tissue and can regulate cellular processes such as chemotaxis, angiogenesis, mitogenesis, differentiation, and metabolism .

Topical retinoids are used in the treatment of both noninflammatory and inflammatory acne.Food and Drug Administration (FDA) approved three topical retinoids: adapalene, tazarotene, and tretinoin. These agents help normalize follicular keratinization and decrease keratinocyte cohesiveness, thereby reducing follicular occlusion and comedon formation .Topical retinoids also compete with factors involved in the acne inflammation response, enhance penetration of other topical acne medications, and accelerate the resolution of acne-induced post-inflammatory hyperpigmentation.

Updates from the Global Alliance on Improving Outcomes in Acne consider topical retinoids as first-line therapy, individually or in combination with benzoyl peroxide. However, the common side effects of skin irritation and discomfort may impede adherence to long-term therapy.

For patients with acne, combination therapy with a topical retinoid and platelet-rich plasma (PRP) has not yet been tested.

PRP with topical retinoids will be evaluated and campared with topical retinoids alone in acne tretment.

ELIGIBILITY:
Inclusion Criteria:

* Patients with facial acne vulgaris
* Age from 12 to 35 years old

Exclusion Criteria:

* Pregnant or lactating women.
* patients with history of coagulation disorders.
* chronic diseases (chronic renal failure, hepatic insufficiency, cardiovascular disorders, uncontrolled diabetes mellitus, thyroid disorders, anemia, autoimmune diseases).
* patients with unrealistic expectations.
* Patients received any systemic treatment in the last 6 months.

Ages: 12 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
change of acne lasions | after 1 month of treatment completion
  record percentage of improvement for each patient after completion of the treatment by comparing before and after digital photographs according to quartile grading scale

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No